CLINICAL TRIAL: NCT05234424
Title: Flow Rate Impact on Arterial Carbon Dioxide Accumulation During Transnasal Humidified Rapid-insufflation Ventilation Exchange: a Randomized Cross-over Study
Brief Title: Flow Rate Impact on Arterial Carbon Dioxide During THRIVE
Acronym: ThriVent
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Futility. Inclusion and logistics of study in a clinical situation proved too difficult to continue.
Sponsor: Uppsala University Hospital (Other)
Responsible Party: Principal Investigator, Peter Frykholm, Consultant and Senior Lecturer, Section of Paediatric Anaesthesia and Intensive Care, Uppsala University Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Frykholm2201
Record Dates: First submitted 2022-01-31; First posted 2022-02-10 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Apneic Oxygenation
Keywords: THRIVE; Apneic oxygenation; General anesthesia
MeSH Terms: interventions — Nicotine

STUDY DESIGN:
Intervention Model Description: After induction of general anesthesia, confirmation of adequate face mask ventilation, and successful arterial cannulation, participants will be assigned to THRIVE flow rates in a randomized order.
Who Masked: Participant
Masking Description: The participants are aware of the intervention used, but not aware of the order of flow rate tests.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- THRIVE 40 L/min (Active Comparator): 40 L/min with 100% oxygen for 10 minutes.
  Interventions: Other: THRIVE
- THRIVE 100 L/min (Experimental): 100 L/min with 100% oxygen for 10 minutes.
  Interventions: Other: THRIVE

INTERVENTIONS:
Other: THRIVE — During general anesthesia, apneic oxygenation with a high flow nasal oxygen system is applied for 10 minutes. Video laryngoscopy will be performed to achieve similar airway patency.

SUMMARY:
Apneic oxygenation describes the process of continuous oxygenation of the blood without breathing efforts. This anesthesia technique has been described in the literature for more than 100 years and is sometimes used under general anesthesia, e.g. during surgery of the vocal chords. Although this technique usually provides marked prolongation of the apneic period because of excellent oxygenation, it is limited by the absence of ventilation and the corresponding accumulation of carbon dioxide in the blood. This will lead to worsening respiratory acidosis and associated complications, such as cardiac arrythmias.

In 2015 it was reported that apneic oxygenation with high-flow nasal oxygen delivery systems (HFNO), a device that provides heated humidified oxygen at high flow rates (usually 30-70 L/min), resulted in less carbon dioxide accumulation compared with historical controls. This specific technique of apneic oxygenation was termed transnasal humidified rapid-insufflation ventilation exchange (THRIVE). To date, the impact on different flow rates on blood carbon dioxide accumulation during THRIVE is unknown. Specifically, very high flow rates, exceeding 70 L/min have not been investigated. Therefore, the aim of this trial is therefore to study the rate of accumulation of carbon dioxide during THRIVE at two different flow rates: 40 and 100 L/min.

DETAILED DESCRIPTION:
Eligible participants with signed informed consent presenting for elective surgery will have standard monitoring with ECG, pulse oximetry, blood pressure, train-of-four monitoring and capnography applied at arrival to the operating room. In addition, a circumferential electric impedance tomography thoracic elastic band with equally spaced electrodes will be placed in the 4th to 6th intercostal space. After induction of general anesthesia with a target controlled infusion of Propofol+Remifentanil and muscle relaxation with Rocuronium bromide, adequate face mask ventilation will be confirmed and arterial cannulation will be performed.

Patients will thereafter receive THRIVE at two flow rates for 10 minutes each in a randomized order. During THRIVE, video laryngoscopy will be performed with a grade 2B visualization of the larynx to establish similar airway patency during the interventions.

Before each flow, an end-tidal oxygen value of >0.85 and end-tidal carbon dioxide value of 4.5-5.0 kPa is achieved by controlled pressure regulated volume control ventilation to establish similar arterial partial pressure of oxygen and carbon dioxide at baseline. An arterial blood gas will also be analyzed before the start of each flow rate to ensure that the initial pCO2 is less than 6.0 kPa. Furthermore, a standardized lung recruitment maneuver will be performed to establish similar baseline compliance of the respiratory system.

Termination criteria will be:

* All flow rates have been applied.
* Severe acidemia (pH<7.10), hypercapnia (pCO2>11.0) or desaturation to SpO2 less than 90% for more than 10 seconds. These termination criteria will apply only to the current flow rate being tested. The participant will be mask ventilated until baseline parameters are established and the next THRIVE flow rate according to randomization will be applied.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting for elective surgery

Exclusion Criteria:

* Age <18 or >65 years
* Body Mass Index (BMI) >35 kg m-2
* American Society of Anesthesiology classification > 2
* Physical activity level less than 5 metabolic equivalents
* Obstruction of the upper airways
* Known or high clinical suspicion of difficult airway
* Obstructive sleep apnea syndrome
* Increased risk of aspiration
* Pulmonary or cardiac condition resulting in a reduction of physical activity level equivalent to the New York Heart Association class of 2 or higher.
* Any contraindication to high-flow nasal oxygen therapy or hypercapnia
* Pregnancy or breastfeeding
* Allergy to any of the anesthetic agents used in the study
* Inability to comprehend oral or written information.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-02-08 (Actual); Primary Completion 2024-05-13 (Actual); Study Completion 2024-05-13 (Actual)

PRIMARY OUTCOMES:
Arterial partial pressure of carbon dioxide (PaCO2) accumulation rate | 10 minutes
  Linear mean accumulation rate of PaCO2 during THRIVE (kPa/min)

SECONDARY OUTCOMES:
Arterial partial pressure of oxygen (PaO2) | 10 minutes
  Change of PaO2
Peripheral saturation (SpO2) | 10 minutes
  Change of SpO2 and lowest SpO2
End-tidal carbon dioxide fraction (EtCO2) | 10 minutes
  Change of EtCO2
End-tidal oxygen fraction. (EtO2) | 10 minutes
  Change of EtO2
End-expiratory lung impedance (EELI) | 10 minutes
  Change of EELI measured with electric impedance tomography
Respiratory compliance | 10 minutes
  Change of dynamic and static respiratory compliance
Heart rate | 10 minutes
  Change of heart rate
Blood pressure | 10 minutes
  Change of systolic, diastolic and mean arterial blood pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Frykholm, MD, PhD, Principal Investigator — Uppsala University
Locations (1):
- Uppsala University Hospital, Uppsala, Uppsala County, Sweden

IPD SHARING:
Plan to Share IPD: No